CLINICAL TRIAL: NCT06336837
Title: False Positive Peripheral Blood Culture in Children With Leukaemia: A Prevalence Study
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, SEDA ARDAHAN SEVGİLİ, Assistant Professor, Ege University
Other Study IDs: 24-3T/48
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Nurse's Role; Leukemia
Keywords: blood cultures; contamination; nurses
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Peripheral blood culture bottles
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No arm used.

SUMMARY:
Chemotherapy, the main treatment for childhood leukemia, has side effects on healthy cells. One of the most important of these side effects is the risk of infection due to neutropenia. In clinics, blood culture is the gold standard for the detection of possible infection risk (bacteremia, fungemia, etc.). During the diagnosis and treatment process in children with leukemia, a large number of peripheral or catheter blood cultures are performed. When the culture results are positive, it is accepted that the infection has grown. In some cases, a positive peripheral blood culture result may not be clinically significant. An agent belonging to the skin flora of the patient or the healthcare professional taking the field culture may also cause the blood culture result to be positive. This is called contamination or false positive blood culture. Contaminated cultures may cause prolonged hospitalization, additional medical interventions, unnecessary initiation of antibiotic treatment and related antibiotic resistance, toxicity due to additional drugs and an increase in hospital costs. The peripheral blood culture contamination rate, which is accepted as a quality indicator in some countries, should be below 3%.

In this context, this study aimed to determine the prevalence of false positive peripheral blood cultures by examining the peripheral blood culture results obtained during routine follow-ups from children hospitalized with leukemia in the pediatric hematology clinic. The data will be collected retrospectively covering three years before March 2024 when the ethics committee approval was obtained. Since the relevant clinic cares for approximately 25 new children diagnosed with leukemia annually, the study sample is planned as 75 cases.

DETAILED DESCRIPTION:
A positive peripheral blood culture does not always mean that the individual has a systemic infection. In some cases, a positive blood culture result may also be seen in the event of contamination with the skin flora of the person receiving/receiving the culture. This is called a false positive blood culture. This situation is characterised as a situation that reduces the reliability of the test. Contaminated false positive blood culture is a single culture bottle containing microorganisms belonging to the skin flora (Coagulase Negative Staphylococcus [Staphylococcus epidermidis, Staphylococcus hominis, Staphylococcus capitis, Staphylococcus haemolyticus], Viridans streptococci, Aerococcus, Micrococcus, Propionibacterium spp, Bacillus spp., [except B. Anthracis], Corynebacterium spp. and alpha-gamma haemolytic streptococci, Dermabacter spp., Rothia spp. and Kocuria spp.)

In cases where bacteria grow in blood culture media, it is necessary to distinguish between local skin flora and true pathogenic bacteria. Contaminated culture results in prolonged hospital stay, additional tests, unnecessary exposure of the patient to antimicrobial agents and increased risk of other complications (qualitative change in microorganisms, increased colonisation rates with drug-resistant organisms such as VRE and MRSA, increased Clostridium difficile infection rates). Inappropriate antibiotherapies initiated due to contaminated blood culture results may cause toxic side effects in the patient. One of the most serious negative effects of inappropriately used antibiotics is the development of antibiotic resistance. Due to the large-scale use of inappropriate antibiotics in hospitals, nosocomial flora undergoes a change. This change leads to the disappearance of susceptible microorganisms in the flora and the increase in resistant strains.

In this context, the aim of this study was to determine the prevalence of false positive peripheral blood cultures by retrospectively examining the peripheral blood culture results obtained during routine follow-up from children hospitalised with leukaemia in the paediatric haematology clinic.

Type of Research Quantitative | Descriptive | Archive Search

Population and Sample The population of the research will consist of children who received chemotherapy due to leukemia treatment and whose peripheral blood culture was taken during routine treatment. The sample will consist of pediatric patients who were hospitalized in the Hematology Department Clinic of Ege University Faculty of Medicine Children's Hospital between March 2021 and March 2024 (after the approval of the Ethics Committee, retrospectively from the month of approval (3 years)). Since the number of inpatient cases diagnosed with leukemia in the Pediatric Hematology Clinic is approximately 25 cases per year, it is planned to examine the peripheral blood culture results of 75 different cases in three years.

ELIGIBILITY:
Inclusion Criteria:

* within the time interval of the study being a patient between the ages of 0-18,
* not having any other disease other than leukaemia,
* having received inpatient chemotherapy treatment in PHO
* having a peripheral blood culture test taken from the patient,
* the patient's culture results being accessible through the hospital information system.

Exclusion Criteria:

* the patient was hospitalised in the clinic outside the time frame of the study,
* a diagnosis other than leukaemia
* peripheral blood culture was not taken from the patient or the results could not be accessed through the hospital information system

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children in the 0-18 age group who have been treated for leukaemia as inpatients in the paediatric hermatology oncology clinic and from whom peripheral blood culture was taken for any reason will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
blood culture contamination rate | three year period
  false positive peripheral blood culture

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)